CLINICAL TRIAL: NCT04410562
Title: Hydroxychloroquine Efficacy and Safety in Preventing SARS-CoV-2 Infection and COVID-19 Disease Severity During Pregnancy and Postpartum
Acronym: COVID-Preg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Barcelona Institute for Global Health (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); University Hospital of Torrejon (Other); Fundación de investigación HM (Other); Hospital Sant Joan de Deu (Other); Hospital del Mar (Other); Hospital Universitario Infanta Leonor (Other); Hospital Universitario Fundación Alcorcón (Other); Hospital General de Segovia (Other); Institut Català de la Salut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-001587-29
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-04

CONDITIONS: Pregnancy Related; COVID; Covid-19
Keywords: pregnancy; covid-19; coronavirus; hydroxychloroquine
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled multicentre clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Experimental): Participants will be then randomized in a 1:1 ratio to HCQ (400 mg/day for three days, followed by 200 mg/day for 11 days)
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Participants will be then randomized in a 1:1 ratio to placebo (2 tablets for three days, followed by one tablet for 11 days).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Participants will receive a bottle containing 19 tablets of study medication. They will be instructed to take two tablets for the first three days and one tablet for the following 11 days. (400 mg/day for three days, followed by 200 mg/day for 11 days).
  Other Names: Dolquine
  Arms: Hydroxychloroquine
Drug: Placebo — Participants will receive a bottle containing 19 tablets of placebo. They will be instructed to take two tablets for the first three days and one tablet for the following 11 days.
  Arms: Placebo

SUMMARY:
It still unclear how SARS-CoV-2 affects pregnant women and their offspring, as well as which factors may influence obstetrical disease and outcomes, including the timing of maternal viral exposure by gestational age, the effects of parity, age, host immune responses, coexisting medical and obstetrical conditions and the effects of treatment regimens. While further information is gathered, based on the existing evidence from other infections causing pneumonia, pregnant women should be considered to be at high risk for developing severe infection during the current COVID-19 epidemic. Results from clinical trials with HCQ in nonpregnant adults may not be directly extrapolated to pregnant women given the special features of the pregnancy status. Thus, clinical research is urgently needed to improve the care and reduce the risk of poor pregnancy outcomes of women in this and in future epidemics.

DETAILED DESCRIPTION:
This is a randomized, double blinded, placebo-controlled multicenter clinical trial including 714 pregnant women (200 SARS-CoV-2 infected -100 symptomatic with mild disease and 100 asymptomatic- pregnant women and 514 SARS-CoV-2 uninfected pregnant women who are contacts with a SARS-CoV-2 case) with the main objectives of assessing the safety and efficacy of oral hydroxychloroquine (HCQ) in reducing maternal viral shedding by PCR, and preventing incident SARS-CoV-2 infection and disease severity. Pregnant women undergoing antenatal follow up at five maternity hospitals, presenting at least one sign and/or one mild suggestive symptoms and a positive SARS-CoV-2 PCR test, or who are contacts of a suspected or confirmed case, will be recruited and randomized 1:1 to receive HCQ orally (400 mg/day for 3 days, followed by 200 mg/day for 11 days) or placebo. Women will be followed up for the duration of the intervention. One week after intervention completion, a SARS-CoV-2 PCR test will be repeated. At delivery, the pregnancy outcome will be registered, and a cord blood sample will be collected to measure for IgG and IgM of SARS-CoV-2. A neonatal nasopharyngeal aspirate will be collected to perform PCR SARS-CoV-2 testing.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with fever (≥37.5ºC) and/or one mild symptom suggestive of COVID-19 disease (cough, dyspnoea, chills, odynophagia, diarrhoea, muscle pain, anosmia, taste disorder, headache) OR contact of a SARS-CoV-2 confirmed or suspected case in the past 14 days
* More than 12 weeks of gestation (dated by ultrasonography)
* Agreement to deliver in the study hospitals

Exclusion Criteria:

* Known hypersensitivity to HCQ or other 4-aminoquinoline compounds
* History of retinopathy of any aetiology
* Concomitant use of digoxin, cyclosporine, cimetidine
* Known liver disease
* Clinical history of cardiac pathology including known long QT syndrome
* Unable to cooperate with the requirements of the study
* Participating in other intervention studies
* Delivery onset (characterized by painful uterine contractions and variable changes of the cervix, including some degree of effacement and slower progression of dilatation up to 5 cm for first and subsequent labours)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Number of PCR confirmed cases among pregnant women | 21 days after intervention
  Number of PCR-confirmed infected pregnant women assessed from collected nasopharyngeal and oropharyngeal swabs at day 21 after treatment start

SECONDARY OUTCOMES:
Incidence of COVID-19 disease during pregnancy | through study completion, an average of 1 year
Incidence of COVID-19-related admissions | through study completion, an average of 1 year
Incidence of all-cause admissions | through study completion, an average of 1 year
Incidence of all-cause outpatient attendances | through study completion, an average of 1 year
Mean duration of symptoms-signs of COVID-19 | through study completion, an average of 1 year
Frequency and severity of adverse events | through study completion, an average of 1 year
Incidence of preeclampsia | through study completion, an average of 1 year
Incidence of gestational diabetes | through study completion, an average of 1 year
Incidence of SARS-CoV-2 infections during pregnancy | through study completion, an average of 1 year
Prevalence of intrauterine growth restriction | through study completion, an average of 1 year
Maternal mortality rate | through study completion, an average of 1 year
Proportion of neonates with SARS-CoV-2- intrauterine infection by PCR-confirmed SARS-CoV-2-infection in nasopharyngeal aspirate. | through study completion, an average of 1 year
Proportion of neonates with clinical signs/symptoms of COVID-19 | through study completion, an average of 1 year
Prevalence of low birth weight (<10th centile according to local standards) | through study completion, an average of 1 year
Prevalence of preterm birth (<37 weeks of gestational age) | through study completion, an average of 1 year
Prevalence of embryo and foetal losses (miscarriages and stillbirths) | through study completion, an average of 1 year
Frequency of congenital malformations | through study completion, an average of 1 year
Proportion of adverse perinatal outcome | through study completion, an average of 1 year
Neonatal morbidity | through study completion, an average of 1 year
Neonatal mortality rate | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital General de Segovia, Segovia, Cartilla Y León
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Clínic de Barcelona, Barcelona, Catalonia
  - Hospital de la Sant Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Catalonia
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - HM Puerta del Sur, Móstoles, Madrid
  - Hospital Universitario de Torrejón, Torrejón de Ardoz, Madrid
  - Hospital Universitario Infanta Leonor, Madrid

IPD SHARING:
Plan to Share IPD: Yes
It would be shared at time of publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: By the end of study

REFERENCES:
- [Derived] Gonzalez R, Gonce A, Gil MDM, Mazarico E, Ferriols-Perez E, Toro P, Llurba E, Saez E, Rodriguez-Zambrano MA, Garcia-Otero L, Lopez M, Santacruz B, Roman MA, Paya A, Alonso S, Cruz-Lemini M, Pons-Duran C, Herrera LB, Chen H, Bardaji A, Quinto L, Menendez C; COVID-Preg research group. Efficacy and safety of hydroxychloroquine for treatment of mild SARS-CoV-2 infection and prevention of COVID-19 severity in pregnant and postpartum women: A randomized, double-blind, placebo-controlled trial. Acta Obstet Gynecol Scand. 2024 Mar;103(3):602-610. doi: 10.1111/aogs.14745. Epub 2023 Dec 14. PMID 38098221
- [Derived] Gonzalez R, Garcia-Otero L, Pons-Duran C, Marban-Castro E, Gonce A, Llurba E, Gil MDM, Rodriguez-Zambrano MA, Chen H, Ramirez M, Bardaji A, Menendez C. Hydroxychloroquine efficacy and safety in preventing SARS-CoV-2 infection and COVID-19 disease severity during pregnancy (COVID-Preg): a structured summary of a study protocol for a randomised placebo controlled trial. Trials. 2020 Jul 2;21(1):607. doi: 10.1186/s13063-020-04557-y. PMID 32616063